CLINICAL TRIAL: NCT02135237
Title: Contingency Management for Alcohol Use Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Sheila Alessi, Associate Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-204H-2; R01AA021446 (NIH)
Record Dates: First submitted 2014-02-24; First posted 2014-05-09 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Alcohol Use Disorder; Contingency Management
MeSH Terms: conditions — Alcoholism | interventions — Ethanol; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Standard Care
  Interventions: Behavioral: Standard Care
- Experimental Group (Experimental): Standard Care plus Prize Contingency Management for Alcohol Abstinence
  Interventions: Behavioral: Prize Contingency Management for Alcohol Abstinence; Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Prize Contingency Management for Alcohol Abstinence — The systematic reinforcement of desired behaviors and the withholding of reinforcement for undesired behaviors
  Arms: Experimental Group
Behavioral: Standard Care

SUMMARY:
Contingency management (CM) treatments are highly efficacious in improving outcomes of substance abusing patients. However, CM has rarely been applied to individuals with alcohol use disorders, primarily because of technological limitations in monitoring drinking. The Secure Continuous Remote Alcohol Monitor (SCRAMx®) is a new technology designed to continuously monitor alcohol consumption 24 hours a day for 7 days per week. The purpose of this study is to evaluate the efficacy of CM in reducing alcohol use using SCRAMx. In total, 120 alcohol abusing or dependent patients initiating outpatient treatment at community-based clinics will be randomly assigned to one of two conditions: standard care, or standard care plus CM with reinforcement based on results of SCRAMx readings. Compared with standard care, it is expected that CM will result in fewer drinking days and longer durations of continuous non-drinking days.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* current diagnosis of alcohol use disorder and self report of recent alcohol use
* pass an informed consent quiz
* agree to wear a SCRAMx monitor for 12 weeks
* have a standard SCRAMx compatible phone line in their home or agree to attend the clinic weekly for brief research visits/downloads
* agree to sign an off-campus property transfer form and return SCRAMx equipment

Exclusion Criteria:

* serious, uncontrolled psychiatric illness
* in recovery from pathological gambling
* have an unstable address
* intend to participate in activities incompatible with SCRAMx over the next 3 months
* are wearing SCRAMx for legal purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
longest duration of abstinence from alcohol | three months
  objective report of alcohol use as measured by SCRAMx device

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Alessi, Ph.D., Principal Investigator — UConn Health
Locations (3):
- United States (3):
  - The Hospital of Central Connecticut at New Britain General, New Britain, Connecticut
  - Farrell Treatment Center, New Britain, Connecticut
  - Behavioral Health Network, Inc., Springfield, Massachusetts